CLINICAL TRIAL: NCT02573194
Title: The Acute Effect of Breakfasts Varying in Protein Source Content on Subjective Appetite Ratings and Voluntary Energy Intake in Healthy Subjects
Brief Title: The Effect of Breakfasts Varying in Protein Source on Appetite and Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Anestis Dougkas, Postdoctoral Research Fellow, Lund University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: FHSC
Record Dates: First submitted 2015-10-08; First posted 2015-10-09 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Obesity
Keywords: Appetite; Amino acids; Protein Source
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Animal source of proteins (Experimental): Breakfast based on animal proteins: 1700 kJ, 25 E% Protein Acute effect of breakfasts varying in protein source content on appetite and energy intake
  Interventions: Dietary Supplement: Breakfasts varying in protein source content on appetite
- Plant source of proteins (Experimental): Breakfast based on plant proteins: 1700 kJ, 25 E% Protein Acute effect of breakfasts varying in protein source content on appetite and energy intake
  Interventions: Dietary Supplement: Breakfasts varying in protein source content on appetite
- Animal and plant source of proteins (Experimental): Breakfast based on both animal and plant proteins: 1700 kJ, 25 E% Protein Acute effect of breakfasts varying in protein source content on appetite and energy intake
  Interventions: Dietary Supplement: Breakfasts varying in protein source content on appetite
- Low protein (Experimental): Breakfast very low in protein: 1700 kJ, 5 E% Protein Acute effect of breakfasts varying in protein source content on appetite and energy intake
  Interventions: Dietary Supplement: Breakfasts varying in protein source content on appetite

INTERVENTIONS:
Dietary Supplement: Breakfasts varying in protein source content on appetite — In this randomized, within-subject study, subjects are asked to consume 4 iso-energetic and iso-volumetric puddings as breakfast (20% of estimated energy requirements) with varying distribution of protein sources. The objective is to identify the protein source and the distribution on suppressing appetite.

SUMMARY:
Over the last decades, changes in the diet and lifestyle have led to overall energy imbalance becoming commonplace and the emergence of an obesity epidemic with more than 1.6 billion adults being overweight.

Consumption of foods that can affect appetite by increasing satiety could regulate the total energy intake and thus body weight. There is data suggesting that the macronutrient composition of the foods and especially protein content may have a potent role on satiety. However, the type of protein appears to play a role in satiety possibly due to the different balance of the amino acid profile.

The research project is dedicated to identify the source (animal or plant) and the optimized protein quantity needed to accelerate satiation, suppress appetite and extend satiety until hunger appears again.

It is hypothesized that the consumption of animal derived protein-enriched meals will induce a reduction in hunger through the impact on gut hormones and peptides that are closely related to the short-term regulation of food intake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Age range 18-50 years
* Normal weight and overweight people as classified by BMI:20-29.9 kg/m2 (inclusive).
* Weight stable (within 3 kg) two months prior to study inclusion
* Understanding English well and feeling comfortable speaking it

Exclusion Criteria:

* Dietary protein consumption >25% energy from protein
* Had surgery in the previous 12 months
* Have suffered a myocardial infarction or stroke at any time
* Suffer from any blood-clotting disorder or prescription of any medication affecting blood clotting
* Suffer from any metabolic disorders (e.g. diabetes, metabolic syndrome or hypertension)
* Any requirement to take long-term medication, especially those active on the gastro-intestinal tract or for cardio-vascular disease
* Any dietary restrictions or recently/currently on a weight reducing diet
* Irregular eating patterns or not regularly consuming breakfast
* Food allergies (e.g. milk protein allergies) or intolerances (e.g. lactose)
* Use of medication which affects food intake or behaviour (e.g. anti-depressants)
* Use of medication likely to affect taste, smell or appetite
* Eating restraint based on the three Factor Eating Questionnaire
* Use of any protein supplements
* A history of alcohol or drug misuse (the average daily number of units of alcohol considered as acceptable is 2-3 units women; 3-4 units men
* Smoking
* Athletes in training (>10 h exercise/week)
* Female that is breast-feeding, pregnant, or if of child-bearing potential and are not using effective contraceptive precautions
* Involvement in a study involving an experimental drug/medication within 3 months prior to entry of this study
* Blood pressure > 160/90 mmHg
* Vegan or Vegetarian
* Glucose > 6 mmol/L
* Gamma glutamyl transpeptidase (liver enzymes) > 1.9 μkat / L
* Alanine aminotransferase > 1.1 μkat / L
* Cholesterol > 6.5 mmol/L
* Triglycerides > 2.0 mmol/L

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in perceived appetite and satiety | Assessed every 30 min for 240 min and 60 min throughout the day after each of the four breakfasts which are served at least one week apart (4 weeks)
  The appetite profile is assessed using validated Visual Analogue Scales (VAS) ratings (i.e hunger, fullness, desire to eat, prospective food consumption). The Questionnaires are performed electronically in personal laptops using the Adaptive Visual Analogue Scales (AVAS) software until 240min and in paper form throughout the remaining of the study day.

SECONDARY OUTCOMES:
Voluntary energy intake | Energy intake is assessed 210 min after the 4 test breakfasts, which are served one week apart.]
  Energy intake is assessed by voluntary hot meal ('Pytt I Panna', Swedish hash) provided 210 min after the test puddings, which are given as breakfast. Subjects are instructed to eat only until they feel comfortable satisfied and are given 25min to consume the meal. The total energy consumed is monitored.
Appetite and Satiety Hormones | Assessed at 6 points in time over the morning of each of the 4 test days, which are separated by 1 week (4 weeks)]
  Blood samples (2 ml) are collected into edetic acid (EDTA) treated tubes at 0 min (fasted blood sample), 30, 60, 90, 150 and 205 min (i.e. total of 6 samples) over the morning on each test day (separated by 1 week) to quantify the plasma concentrations of circulating appetite regulating hormones and amino acids. Protease inhibitors are added to the samples to reduce protein degradation. All samples are centrifuged at 4 C for 10 min at 2000 g after collection and are separated and stored in cryogenic vials at -80 C.
Hedonic Ratings and Palatability of the Test Breakfasts and Meals | Assessed immediately after consumption of the 4 test puddings and Swedish hash meal (4 weeks)
  The palatability and hedonic ratings are assessed using validated Visual Analogue Scales (VAS) ratings (i.e appearance, taste, overall palatability). The Questionnaires are performed electronically in personal laptops using the Adaptive Visual Analogue Scales (AVAS) software.
Glucose measurements | Assessed at 7 points in time over the morning of each of the 4 test days, which are separated by 1 week (4 weeks)
  Capillary blood samples are collected by finger-prick at 0 min (fasted blood sample), 30, 45, 60, 90, 150 and 205 min (i.e. total of 7 samples) over the morning on each test day (separated by 1 week) to quantify the glucose concentration using HemoCue Glucose System.

CONTACTS AND LOCATIONS:
Overall Officials: Anestis Dougkas, PhD, Principal Investigator — Lund University
Locations (1):
- Food for Health Science Center, Lund, Skåne County, Sweden